CLINICAL TRIAL: NCT00714909
Title: CAVECCAS Value of Risk Factors for Symptomatic Catheter Related Thrombosis in Patients With Breast Cancer Treated With Adjuvant Chemotherapy
Brief Title: Determination of Predictive Value of Echography Doppler Abnormalities
Acronym: CAVECCAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle Brindel, Department Clinical Research of developpement
Other Study IDs: K070104
Record Dates: First submitted 2008-07-11; First posted 2008-07-14 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer; Upper Extremity Deep Vein Thrombosis, Secondary
Keywords: Breast cancer; Catheter related thrombosis; Diagnosis; Echography doppler; Risk factors
MeSH Terms: conditions — Breast Neoplasms; Upper Extremity Deep Vein Thrombosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
In order to avoid to use a traumatic and iatrogenic examen (phlebography), the purpose of the study is to validate echography doppler in the diagnosis of asymptomatic related catheter related thrombosis.

DETAILED DESCRIPTION:
Phlebography is the gold standard for the diagnosis of asymptomatic catheter related thrombosis but can not be performed in about 15% of patients because of arm swelling and lack of superficial veins.

Echography doppler is an easy, cheap and atraumatic way to make the diagnosis of deep vein thrombosis. The value of echography doppler has been proven for the diagnosis of symptomatic deep venous thrombosis of lower and upper limbs and for the diagnosis of proximal asymptomatic lower limbs.

To validate the echography doppler we intend to correlate asymptomatic findings to the occurrence symptomatic related catheter related thrombosis.

Patients with localized breast cancer treated with chemotherapy will be enrolled in the study. An echography doppler will be performed on day 8, 30 and 90 after catheter insertion. Findings in asymptomatic patients (thrombus visualisation, lack of vein compressibility, variation of physiologic vein blood flow) will thereafter be correlated with the presence or absence of clinical signs of catheter related thrombosis.

In order to assess if they are risk factors for catheter related thrombosis, we will determine the level D-Dimer, microparticles and the results of generation thrombin tests before and 2 days after catheter insertion.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* histologically proven breast cancer
* localized breast cancer without metastasis
* adjuvant or neo adjuvant chemotherapy
* insertion of central catheter with port for chemotherapy
* central catheter for more than three months
* inform consent
* follow up for three months

Exclusion Criteria:

* ongoing anticoagulant therapy
* previous central catheter
* femoral catheter
* double lumen catheter
* central catheter without port
* platelets < 80G/L, TQ < 50%, fibrinogen < 1 g/L
* creatinin > 175mole/L

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated receiving adjuvant chemotherapy for localized breast cancer in the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Symptomatic catheter related thrombosis, as confirmed by echography doppler, phlebography or angiography scan | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe M Debourdeau, MD, Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (1):
- Saint-Louis Hospital, Paris, France